CLINICAL TRIAL: NCT02411292
Title: Enoxaparin Metabolism in Reconstructive Surgery Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Pannucci, Assistant Professor, Plastic Surgery, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB 00079118
Record Dates: First submitted 2015-03-30; First posted 2015-04-08 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis; Pulmonary Embolus; Reconstructive Surgery
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enoxaparin metabolism (Experimental): Eligible patients will have steady state peak and trough anti-Xa levels drawn after the third enoxaparin dose. For patients in-range (levels 0.3-0.5IUmL), no intervention will be undertaken. For patients out of range, enoxaparin dose will be adjusted according to an established dose adjustment algorithm. Repeat levels will be checked after the third administration of the new dose.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Enrolled patients will receive real-time monitoring of peak and trough steady state anti-Xa levels. Out-of-range patients will receive real time dose adjustment of Enoxaparin using a clinical protocol developed with our inpatient pharmacists.

SUMMARY:
Venous thromboembolism (VTE) is a leading cause of death among hospitalized patients, and is an important patient safety issue in plastic surgery. Previous work has shown that enoxaparin prophylaxis can prevent many post-operative VTE events, and current American Society of Plastic Surgeons guidelines support enoxaparin prophylaxis for high-risk patients. Highest risk patients often have cancer or trauma reconstruction. Primary outcomes include 1) peak and trough steady-state aFXa levels in response to standard and escalated doses of enoxaparin and 2) the proportion of patients with appropriate aFXa levels pre and post initiation of a clinical protocol for enoxaparin dose adjustment. The investigators expect that standard dosing will result in inadequate aFXa peak and trough levels, and that the clinical dose adjustment protocol will significantly improve the proportion of in-range aFXa levels. The investigators will also develop a linear regression-based equation to calculate, based on patient-level factors, the required dose of enoxaparin to generate in-range aFXa levels. This research may show that the current "one size fits all" approach to enoxaparin prophylaxis is insufficient. In the trauma and orthopaedic populations, patients with low initial aFXa levels are significantly more likely to develop deep venous thrombosis. Thus, this study has important implications for appropriate enoxaparin dose magnitude and frequency, and may ultimately help to decrease the substantial morbidity and mortality associated with post-operative VTE.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a leading cause of death among hospitalized patients, and is an important patient safety issue in plastic surgery. Previous work has shown that enoxaparin prophylaxis can prevent many post-operative VTE events, and current American Society of Plastic Surgeons guidelines support enoxaparin prophylaxis for high-risk patients. However, the Plastic Surgery Foundation-funded Venous Thromboembolism Prevention Study showed that 1 in 25 highest risk patients still had a "breakthrough" VTE event despite receipt of guideline-compliant enoxaparin prophylaxis. Highest risk patients often have cancer or trauma reconstruction. These surgeries may have surgical injury that is equal in scope to patients with traumatic or thermal injury. Previous work in patients with traumatic or thermal injury has shown that enoxaparin metabolism, measured by anti-factor Xa (aFXa) level, is substantially increased: a higher degree of injury is associated with higher enoxaparin dose requirements to achieve prophylactic levels. "Breakthrough" VTE events may occur in plastic and reconstructive surgery patients due to inadequate enoxaparin dosing. The investigators will examine enoxaparin pharmacokinetics and test whether a clinical protocol for real-time enoxaparin dose adjustment can favorably alter the proportion of patients with in-range aFXa levels. Primary outcomes include 1) peak and trough steady-state aFXa levels in response to standard and escalated doses of enoxaparin and 2) the proportion of patients with appropriate aFXa levels pre and post initiation of a clinical protocol for enoxaparin dose adjustment. The investigators expect that standard dosing will result in inadequate aFXa peak and trough levels, and that the clinical dose adjustment protocol will significantly improve the proportion of in-range aFXa levels. The investigators will also develop a linear regression-based equation to calculate, based on patient-level factors, the required dose of enoxaparin to generate in-range aFXa levels. This research may show that the current "one size fits all" approach to enoxaparin prophylaxis is insufficient. In the trauma and orthopaedic populations, patients with low initial aFXa levels are significantly more likely to develop deep venous thrombosis. Thus, this study has important implications for appropriate enoxaparin dose magnitude and frequency, and may ultimately help to decrease the substantial morbidity and mortality associated with post-operative VTE.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will include:

* adult (age ≥18) patients presenting for reconstructive surgery under general anesthesia.
* expected post-operative stay will be at least three days to allow peak aFXa levels to be drawn.
* eligible patients will include those having major reconstructive surgery.

Exclusion Criteria:

Exclusion criteria will include:

* contraindication to use of enoxaparin,
* intracranial bleeding/stroke,
* hematoma or bleeding disorder,
* known heparin-induced thrombocytopenia,
* creatinine clearance ≤30mL/min,
* serum creatinine >1.6mg/dL, or epidural anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Puccini, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Paolini G, Firmani G, Sorotos M, Ninkovic M, Santanelli di Pompeo F. European guidelines on peri-operative venous thromboembolism prophylaxis: first update.: Chapter 8: Plastic surgery. Eur J Anaesthesiol. 2024 Aug 1;41(8):598-603. doi: 10.1097/EJA.0000000000001998. Epub 2024 Jul 10. No abstract available. PMID 38957026
- [Derived] Pannucci CJ, Fleming KI, Varghese TK Jr, Stringham J, Huang LC, Pickron TB, Prazak AM, Bertolaccini C, Momeni A. Low Anti-Factor Xa Level Predicts 90-Day Symptomatic Venous Thromboembolism in Surgical Patients Receiving Enoxaparin Prophylaxis: A Pooled Analysis of Eight Clinical Trials. Ann Surg. 2022 Dec 1;276(6):e682-e690. doi: 10.1097/SLA.0000000000004589. Epub 2020 Oct 19. PMID 33086312
- [Derived] Pannucci CJ, Fleming KI, Agarwal J, Rockwell WB, Prazak AM, Momeni A. The Impact of Once- versus Twice-Daily Enoxaparin Prophylaxis on Risk for Venous Thromboembolism and Clinically Relevant Bleeding. Plast Reconstr Surg. 2018 Jul;142(1):239-249. doi: 10.1097/PRS.0000000000004517. PMID 29649055
- [Derived] Pannucci CJ, Fleming KI. Comparison of face-to-face interaction and the electronic medical record for venous thromboembolism risk stratification using the 2005 Caprini score. J Vasc Surg Venous Lymphat Disord. 2018 May;6(3):304-311. doi: 10.1016/j.jvsv.2017.10.016. Epub 2018 Feb 13. PMID 29452956

RESULTS

PARTICIPANT FLOW:
Groups:
- Enoxaparin Metabolism: Eligible patients will have steady state peak and trough anti-Xa levels drawn after the third enoxaparin dose. For patients in-range (levels 0.3-0.5IUmL), no intervention will be undertaken. For patients out of range, enoxaparin dose will be adjusted according to an established dose adjustment algorithm. Repeat levels will be checked after the third administration of the new dose.
  Enoxaparin: Enrolled patients will receive real-time monitoring of peak and trough steady state anti-Xa levels. Out-of-range patients will receive real time dose adjustment using a clinical protocol developed with our inpatient pharmacists.
Period: Overall Study
Arm/Group | Enoxaparin Metabolism
Started | 110
Completed | 89
Not Completed | 21
Not completed — Discharged before 3rd enoxaparin dose | 16
Not completed — Death | 2
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: The sixteen participants that were discharged before the third enoxaparin dose were excluded from the analysis.
Arm/Group | Enoxaparin Metabolism
Number analyzed (Participants) | 94
Age, Continuous [Mean (Full Range); unit: years] | 52.6 [21 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 79
  Ethnicity: African American | 1
  Ethnicity: Native American or Alaskan Native | 4
  Ethnicity: Hispanic or Latino | 9
  Ethnicity: Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 94
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 28.6 [17 to 49.8]
Gross weight [Mean (Full Range); unit: lbs] | 184 [94 to 320]
Number of patients receiving treatment for Diabetes [Count of Participants; unit: Participants] | 8
Creatinine [Mean (Full Range); unit: mg/dL] | 0.82 [0.34 to 1.52]
Current smoker [Count of Participants; unit: Participants] | 14
Caprini Score [Median (Full Range); unit: scores on a scale] — The Caprini risk score is a risk assessment tool for the occurrence of venous thromboembolism (VTE) among surgical patients. The Caprini risk score includes 40 factors, each ascribed points ranging from 1 to 5. The Caprini score is calculated by adding the scores of all factors present in the patient. The minimum possible score is 0. The maximum score for men is 85. The maximum score for women is 88. The Caprini score is interpreted in the following way:
  Score 0-1: Low risk of VTE
  Score 2: Moderate of VTE
  Score 3-4: High risk of VTE
  Score ≥ 5: Highest risk for VTE
  scores on a scale | 7 [2 to 15]
Location of primary operation [Count of Participants; unit: Participants]
  Head and neck | 2
  Breast | 29
  Chest, nonbreast | 5
  Back including pressure ulcers | 26
  Upper extremity | 2
  Lower extremity | 30
Length of operation [Mean (Full Range); unit: minutes] | 281 [23 to 996]
Total body surface area surgically injured [Mean (Full Range); unit: percentage of total body surface area] | 6.1 [1 to 13]
Length of hospital stay [Mean (Full Range); unit: days] | 7.6 [3 to 39]
Length of chemoprophylaxis [Mean (Full Range); unit: days] | 10.3 [1 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Venous Thromboembolism Events
Description: Any symptomatic venous thromboembolism events, including deep venous thrombosis or pulmonary embolus occurring within 90 days of surgery
Time Frame: 90 days
Population: Patients with out-of-range levels or missing levels were dropped from relevant analyses. Of the 89 participants who completed the study, 88 had peak steady-state anti-factor Xa levels to be analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Low aFXa Level: Patients with a low Anti-Factor Xa Level as identified after the third administration of enoxaparin
- In-Range or High aFXa Level: Patients with an in-range or high Anti-Factor Xa Level as identified after the third administration of enoxaparin
Arm/Group | Low aFXa Level | In-Range or High aFXa Level
Number analyzed (Participants) | 49 | 39
Participants | 5 | 0

2. Primary Outcome: Number of Participants With Bleeding Events
Description: Bleeding events requiring alteration in the course of care within 90 days of surgery
Time Frame: 90 days
Population: Bleeding events are reported for the 94 who were not discharged prior to the third Enoxaparin dose. Because two bleeding events occurred prior to the drawing of labs, they cannot be classified into low vs. in-range/high enoxaparin levels. Because of this, reporting on bleeding events is reported across the whole study population and not by arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Enoxaparin Metabolism
Number analyzed (Participants) | 94
Participants | 3

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Enoxaparin Metabolism
All-Cause Mortality (participants affected / at risk) | 2/110
Serious Adverse Events (participants affected / at risk) | 2/110
Other Adverse Events (participants affected / at risk) | 8/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enoxaparin Metabolism (N=110)
Death (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enoxaparin Metabolism (N=110)
Deep venous thrombosis (Vascular disorders) | 4 (4)
Pulmonary Embolism (Vascular disorders) | 1 (1)
Bleeding (Vascular disorders) | 3 (3) — Bleeding events changing the course of care

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes